CLINICAL TRIAL: NCT06347887
Title: Clinical Validation of ColonAiQ (a Blood-based Assay Targeting Circulating Tumor DNA Methylation) for Colorectal Cancer Detection
Brief Title: Clinical Validation of ColonAiQ (a Blood-based Assay Targeting ctDNA Methylation) for Colorectal Cancer Detection
Status: Completed | Type: Observational
Sponsor: Singlera Genomics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SGI-PCR-01
Record Dates: First submitted 2024-03-27; First posted 2024-04-04 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colorectal cancer group: Patients who are 18 years of age and older and diagnosed with colorectal cancer.
  Interventions: Diagnostic Test: ColonAiQ test and Colonoscopy
- Control group: Patients with other non-neoplastic diseases of the digestive system, and patients with non-colorectal cancer such as gastric cancer, esophageal cancer, breast cancer and lung cancer, etc. as well as Individuals without any diseases checked by colonoscopy.
  Interventions: Diagnostic Test: ColonAiQ test and Colonoscopy

INTERVENTIONS:
Diagnostic Test: ColonAiQ test and Colonoscopy — Diagnostic Test

SUMMARY:
The DNA methylation targets in preoperative plasma samples of the subjects will be detected by the multi-gene methylation test (ColonAiQ), and the test accuracy will be evaluated by compared with the clinical diagnosis evidence.

DETAILED DESCRIPTION:
The accuracy of ColonAiQ test in clinical testing will be evaluated in the multicenter, prospective study. Patients with colorectal cancer, intestinal polyps, adenomas and other non-neoplastic diseases of the digestive system, and patients with non-colorectal cancer such as gastric cancer, esophageal cancer, breast cancer and lung cancer will be enrolled. In this study, all cfDNA will be tested by fluorescence quantitative PCR, and some samples will be tested by NGS to verify the effectiveness of ColonAiQ test. Clinical diagnosis reports and methylation test results will be blinded to the lab tester and clinician respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, gender is not limited;
2. meet one of the following conditions: 1) Suspected colorectal cancer (CRC); 2) Diagnosed with CRC according to clinical diagnostic criteria; 3) Do not have CRC and have interfering diseases:

   1. Confirmed non-CRC digestive tract cases: colorectal polyps, adenomas, and other benign diseases of the digestive system;
   2. Confirmed cases of other cancers other than CRC: gastric, esophageal, breast, and lung cancer;
   3. diseases where the same gene methylation may be present (non-rheumatoid arthritis, etc.);
3. The subject or his/her guardian is able to understand the purpose of the study, demonstrate sufficient adherence to the study protocol, and sign the informed consent.

Exclusion Criteria:

1. People who cannot tolerate relevant tests for clinical diagnosis;
2. Pregnant women;
3. Patients who have previously received colorectal cancer surgery, tumor drug therapy, neoadjuvant therapy, or radiotherapy;
4. Other conditions deemed unsuitable for inclusion by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years of age and older who are eligible for colorectal cancer diagnosis and scheduled for a screening colonoscopy. more than 1000 subjects are targeted to enroll.
Sampling Method: Probability Sample
Enrollment: 1965 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Sensitivity for colorectal cancer with ColonAiQ test | Up to 32 months
  The proportion of participants with colorectal cancer who have positive test results
Specificity for colorectal cancer with ColonAiQ test | Up to 32 months
  The proportion of negative test results among participants without CRC and other diseases

SECONDARY OUTCOMES:
PPV for colorectal cancer with ColonAiQ test | Up to 32 months
  Positive Predictive Value: the proportion of positive test participants who are colorectal cancer patients.
NPV for colorectal cancer with ColonAiQ test | Up to 32 months
  Negative Predictive Value: the proportion of negative test participants who have no disease checked by colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Guoxiang Cai, M.D. Ph.D., Principal Investigator — Fudan University
Locations (7):
- China (7):
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Cancer Hospital Affiliated to Shandong First Medical University (Shandong Institute of Cancer Prevention and Control, Shangdong Cancer Hospital), Jinan, Shandong
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Xi'an Daxing Hospital, Xi’an, Shanxi
  - Xi'an Gaoxin Hospital, Xi’an, Shanxi
  - Zhejiang provincial people's hospital, Hangzhou, Zhejiang
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data that underlie the results reported in publications of the study may be shared after de-identification.